CLINICAL TRIAL: NCT00003466
Title: Phase II Treatment of Adults and Children With Progressive Low Grade Gliomas With Temodal
Brief Title: Temozolomide in Treating Patients With Progressive Low-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1703 (CDR0000066502); DUMC-1703-04-12R7; DUMC-000693-01-3R1; DUMC-1703-01-94R; DUMC-1502-97-10; DUMC-1569-98-10R1; DUMC-97125; NCI-G98-1469; DUMC-1703-02-9R5
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult mixed glioma; childhood mixed glioma; adult pilocytic astrocytoma; adult subependymoma; recurrent childhood cerebral astrocytoma; adult brain stem glioma; recurrent childhood brain stem glioma; untreated childhood brain stem glioma; recurrent childhood visual pathway and hypothalamic glioma; untreated childhood visual pathway and hypothalamic glioma; adult oligodendroglioma; adult diffuse astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioma; Astrocytoma; Glioma, Subependymal; Optic Nerve Glioma; Oligodendroglioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well temozolomide works in treating patients with progressive low-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the response rate in patients with progressive low-grade gliomas treated with temozolomide.
* Determine the activity of this drug, in terms of stabilizing growth of progressive low-grade gliomas, in adult patients.

OUTLINE: Patients are stratified by disease type (pilocytic astrocytoma, mixed glioma, well-differentiated oligodendroglioma, and nonbiopsied optic pathway glioma or pontine glioma).

Patients receive temozolomide orally once daily on days 1-5. Courses repeat every 28 days. In the absence of disease progression or unacceptable toxicity, patients may continue with treatment until tumor has remained stable for 12 courses.

Patients are followed every 8-12 weeks for 2 years.

PROJECTED ACCRUAL: A total of 36-100 patients (9-25 per stratum) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed progressive, primary, intracranial, supratentorial, low-grade glioma including:

  * Astrocytoma
  * Oligodendroglioma
  * Mixed glioma
  * Optic pathway glioma*
  * Pontine glioma* NOTE: *Biopsy not required
* Patients with optic pathway glioma must also meet the following criteria:

  * Progressive loss of vision as defined by doubling of octaves
  * Visual acuity loss not explained by other causes
  * Increase in proptosis of greater than 3 mm
  * Increase in diameter of optic nerve of at least 2 mm on neuroimaging
  * Increase in distribution of tumor involving optic tracts or optic radiations as indicated by CT scan or MRI

PATIENT CHARACTERISTICS:

Age:

* 4 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT less than 2.5 times ULN
* Alkaline phosphatase less than 2 times ULN

Renal:

* Creatinine less than 1.5 times ULN
* BUN less than 1.5 times ULN

Other:

* Must be neurologically stable
* No systemic disease
* No acute infection requiring IV antibiotics
* No frequent vomiting
* No other medical condition that would interfere with oral medication (e.g., partial bowel obstruction)
* No other prior or concurrent malignancies except:

  * Surgically cured carcinoma in situ of the cervix
  * Basal or squamous cell skin cancer
* HIV negative
* No AIDS-related illness
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy (growth factors or epoetin alfa)

Chemotherapy:

* At least 6 weeks since prior chemotherapy unless evidence of disease progression
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 6 weeks since prior radiotherapy unless evidence of disease progression
* No concurrent radiotherapy

Surgery:

* At least 3 weeks since prior surgery unless evidence of disease progression
* Recovered from all prior surgery

Other:

* No other concurrent investigational drugs

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 1998-03; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Response rate
Activity of temozolomide

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (2):
- United States (2):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania